CLINICAL TRIAL: NCT00434356
Title: A Multicenter, Phase II, Randomized, Controlled Trial Evaluating the Efficacy and Safety of Sunitinib in Combination With Bevacizumab and Paclitaxel in Previously Untreated Patients With Metastatic Breast Cancer
Brief Title: A Study of Sunitinib in Combination With Bevacizumab and Paclitaxel in Previously Untreated Patients With Metastatic Breast Cancer (SABRE-B)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on data collected, the combination appeared to be poorly tolearated.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Jai Balkissoon, M.D., Study Director, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVF4057g
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Avastin; MBC; Breast Cancer; Sutent
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Sunitinib; Paclitaxel

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab; Drug: sunitinib; Drug: paclitaxel
- 2 (Placebo Comparator)
  Interventions: Drug: bevacizumab; Drug: paclitaxel

INTERVENTIONS:
Drug: bevacizumab — Intravenous repeating dose
Drug: sunitinib — Oral repeating dose
  Arms: 1
Drug: paclitaxel — Intravenous repeating dose

SUMMARY:
This is a multicenter, Phase II, randomized, controlled, open label trial designed to provide a preliminary assessment of the safety and efficacy of sunitinib when combined with bevacizumab and paclitaxel in patients who have not previously received chemotherapy for locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically or cytologically confirmed adenocarcinoma of the breast with measurable or non-measurable locally recurrent or metastatic disease
* Age ≥ 18 years
* Adequate left ventricular function at study entry, defined as an Left Ventricular Ejection Fraction (LVEF) > 50% by either Multi Gated Acquisition(MUGA) scan or Electrocardiogram (ECHO)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Ability and willingness to comply with study and follow-up procedures

Exclusion Criteria:

* Unknown HER2 status or known HER2-positive status
* Prior chemotherapy for locally recurrent or metastatic disease
* Prior hormonal therapy within 2 weeks prior to Day 1
* Prior adjuvant or neoadjuvant taxane chemotherapy within 12 months prior to Day 1
* Prior adjuvant or neoadjuvant non-taxane chemotherapy within 6 months prior to Day 1
* For patients who have received recent radiotherapy, ongoing Grade ≥ 3 acute toxicity
* Patients with brain metastasis on full dose anticoagulation therapy
* Life expectancy of < 12 weeks
* Current, recent (within 4 weeks of Day 1), or planned participation in an experimental drug study
* Inadequate organ function within 28 days prior to Day 1
* Untreated abnormal thyroid function tests
* Uncontrolled serious medical or psychiatric illness
* Active infection requiring IV antibiotics at enrollment or randomization
* History of other malignancies within 5 years prior to Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Class II or greater CHF
* History of myocardial infarction or unstable angina within 12 months prior to Day 1
* History of stroke or transient ischemic attack within 12 months prior to Day 1
* Known central nervous system (CNS) disease except for treated brain metastasis
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1
* History of hemoptysis within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening, as demonstrated by a urine protein/creatinine ratio of ≥ 1.0 at screening
* Known hypersensitivity to any component of bevacizumab or sunitinib
* Pregnancy (positive pregnancy test) or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Balkissoon, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Paclitaxel + Sunitinib: Bevacizumab will be administered at 10 mg/kg by intravenous (IV) infusion every 2 weeks; paclitaxel will be administered at 90 mg/m2 by IV infusion weekly for 3 weeks followed by 1 week of rest; sunitinib will be administered orally at 25 mg/day or 37.5 mg/day for 3 weeks followed by 1 week of rest
- Bevacizumab + Paclitaxel: Bevacizumab will be administered at 10 mg/kg by intravenous (IV) infusion every 2 weeks; paclitaxel will be administered at 90 mg/m2 by IV infusion weekly for 3 weeks followed by 1 week of rest
Period: Overall Study
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Started | 23 | 23
Completed | 0 | 0
Not Completed | 23 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Customized [Number; unit: participants] — Randomized patients
  participants
    < 18 Years | 0 | 0 | 0
    Between 18 and 40 Years | 2 | 5 | 7
    Between 41 and 64 Years | 15 | 17 | 32
    >= 65 Years | 6 | 1 | 7
Age Continuous [Mean (Standard Deviation); unit: years] — Randomized patients
  years | 57.3 (13.3) | 50.8 (11.7) | 54 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Randomized patients
  Participants
    Female | 23 | 23 | 46
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: The best overall response is the best response, per the Response Evaluation Criteria In Solid Tumors (RECIST) criteria, recorded from randomization until disease progression/recurrence (includes both confirmed and unconfirmed responses). Although the original primary outcome was progression-free survival, there was insufficient data available to report on that outcome.
Time Frame: From randomization until disease progression/recurrence (by patient)
Population: Randomized patients with at least one scan available at baseline and post-baseline
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 17 | 18
participants
  Complete Response | 0 | 0
  Partial Response | 12 | 11
  Stable Disease | 3 | 4
  Progressive Disease | 2 | 2
  Unable to Evaluate | 0 | 1
  Missing | 0 | 0

2. Secondary Outcome: Serious Adverse Events (SAEs)
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0. An SAE is defined as an adverse event that results in death, is life threatening, requires hospitalization, results in significant disability, results in birth defect, or is considered a significant medical event by the investigator
Time Frame: 30 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 23 | 23
participants
  Febrile Neutropenia | 2 | 1
  Haemolytic Anaemia | 1 | 0
  Neutropenia | 0 | 1
  Constipation | 1 | 0
  Diarrhoea | 1 | 0
  Gastrointestinal Perforation | 1 | 0
  Haemorrhoids | 1 | 0
  Vomiting | 1 | 0
  Chest Pain | 0 | 2
  Asthenia | 0 | 1
  Anaphylactic Reaction | 1 | 0
  Drug Hypersensitivity | 0 | 1
  Upper Respiratory Tract Infection | 0 | 2
  Cellulitis | 0 | 1
  Pneumonia | 0 | 1
  Tooth Infection | 1 | 0
  Spinal Compression Fracture | 1 | 0
  Dehydration | 1 | 2
  Hypoglycaemi | 0 | 1
  Syncope | 0 | 1
  Pulmonary Embolism | 1 | 1
  Epistaxis | 0 | 1
  Hypoxia | 0 | 1
  Skin Ulcer | 1 | 0

3. Secondary Outcome: Grade ≥ 3 Adverse Events (AEs)
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0. Grading: 1=Mild AE; 2=Moderate AE; 3=Severe AE; 4=Life-threatening or disabling AE; 5=Death related to AE
Time Frame: 30 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 23 | 23
participants
  Neutropenia | 10 | 2
  Leukopenia | 7 | 0
  Febrile Neutropenia | 3 | 1
  Haemolytic Anaemia | 1 | 0
  Lymphopenia | 1 | 0
  Diarrhoea | 4 | 0
  Constipation | 0 | 1
  Nausea | 1 | 0
  Vomiting | 1 | 0
  Gastrointestinal Perforation | 1 | 0
  Haemorrhoids | 1 | 0
  Small Intestinal Obstruction | 1 | 0
  Fatigue | 6 | 2
  Chest Pain | 0 | 2
  Asthenia | 0 | 1
  Mucosal Inflammation | 0 | 1
  Hyperbilirubinaemia | 1 | 0
  Drug Hypersensitivity | 2 | 1
  Anaphylactic Reaction | 1 | 0
  Upper Respiratory Tract Infection | 0 | 2
  Cellulitis | 0 | 1
  Otitis Media | 1 | 0
  Pneumonia | 0 | 1
  Tooth Infection | 1 | 0
  Urinary Tract Infection | 0 | 1
  Spinal Compression Fracture | 1 | 0
  Thermal Burn | 1 | 0
  Haemoglobin Decreased | 0 | 1
  Neutrophil Count Decreased | 0 | 1
  Dehydration | 1 | 2
  Anorexia | 1 | 0
  Hypoglycaemia | 0 | 1
  Neuropathy Peripheral | 1 | 2
  Headache | 1 | 0
  Migraine | 0 | 1
  Syncope | 0 | 1
  Haematuria | 1 | 0
  Epistaxis | 0 | 1
  Pulmonary Embolism | 1 | 1
  Palmar-Plantar Erythrodysaesthesia Syndrome | 0 | 1
  Skin Ulcer | 1 | 0
  Hypertension | 2 | 1

4. Secondary Outcome: Adverse Events Leading to Death
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 30 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 23 | 23
participants | 0 | 0

5. Secondary Outcome: Adverse Events Leading to Sunitinib Discontinuation, Dose Interruption, or Dose Reduction
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 30 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib
Number analyzed (Participants) | 23
participants
  Neutropenia | 11
  Leukopenia | 6
  Febrile Neutropenia | 2
  Thrombocytopenia | 2
  Lymphopenia | 1
  Diarrhoea | 4
  Nausea | 2
  Vomiting | 2
  Constipation | 1
  Gastrointestinal Perforation | 1
  Haemorrhoids | 1
  Hyperbilirubinaemia | 1
  Anaphylactic Reaction | 1
  Drug Hypersensitivity | 1
  Otitis Media | 1
  Tooth Infection | 1
  Spinal Compression Fracture | 1
  Thermal Burn | 1
  Anorexia | 1
  Dehydration | 1
  Neuropathy Peripheral | 1
  Haematuria | 1
  Skin Ulcer | 1
  Hypertension | 2

6. Secondary Outcome: Adverse Events Leading to Bevacizumab Discontinuation or Dose Interruption
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 30 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 23 | 23
participants
  Neutropenia | 9 | 4
  Leukopenia | 4 | 0
  Febrile Neutropenia | 2 | 0
  Haemolytic Anaemia | 1 | 0
  Lymphopenia | 1 | 0
  Thrombocytopenia | 1 | 0
  Diarrhoea | 3 | 0
  Constipation | 1 | 0
  Gastrointestinal Perforation | 1 | 0
  Gingival Bleeding | 1 | 0
  Nausea | 1 | 0
  Small Intestinal Obstruction | 1 | 0
  Toothache | 0 | 1
  Vomiting | 1 | 0
  Fatigue | 3 | 3
  Chest Pain | 0 | 1
  Mucosal Inflammation | 0 | 1
  Hyperbilirubinaemia | 1 | 0
  Anaphylactic Reaction | 1 | 0
  Otitis Media | 1 | 0
  Pneumonia | 0 | 1
  Rhinitis | 1 | 0
  Skin Infection | 1 | 0
  Upper Respiratory Tract Infection | 0 | 1
  Thermal Burn | 1 | 0
  Dehydration | 1 | 2
  Anorexia | 1 | 1
  Hypoglycaemia | 0 | 1
  Neuropathy Peripheral | 1 | 1
  Memory Impairment | 1 | 0
  Migraine | 0 | 1
  Confusional State | 1 | 0
  Haematuria | 1 | 0
  Proteinuria | 1 | 0
  Epistaxis | 1 | 1
  Dyspnoea | 0 | 1
  Haemoptysis | 0 | 1
  Pulmonary Embolism | 0 | 1
  Dermatitis | 0 | 1
  Skin Ulcer | 1 | 0
  Hypertension | 1 | 0

ADVERSE EVENTS:
Arm/Group | Bevacizumab + Paclitaxel + Sunitinib | Bevacizumab + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 10/23 | 9/23
Other Adverse Events (participants affected / at risk) | 21/23 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Sunitinib (N=23) | Bevacizumab + Paclitaxel (N=23)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hemolytic Anemia (Blood and lymphatic system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforatioin (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Cellulitis (Immune system disorders) | 0 | 1
Tooth Infection (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Paclitaxel + Sunitinib (N=23) | Bevacizumab + Paclitaxel (N=23)
Neutropenia (Blood and lymphatic system disorders) | 13 | 5
Leukopenia (Blood and lymphatic system disorders) | 7 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 8 | 5
Neuropathy Peripheral (Nervous system disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Hemoglobin Decreased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-Plantar Erythrodysasthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Oral Discomfort (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Weight Decreased (Investigations) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Based on the early safety results from this study, further recruitment and treatment was halted. Insufficient efficacy data were available to perform all protocol-specified analyses and limited the interpretation of the analyses performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study.